CLINICAL TRIAL: NCT06855485
Title: A Prospective Single-Center Observational Study on the Evaluation of Efficacy and Safety of HANAROSTEN® HOT Plumber™ With Z-EUSIT™ for Pancreatic Pseudocysts Drainage
Brief Title: Efficacy and Safety of HANAROSTEN® HOT Plumber™ With Z-EUSIT™ for Pancreatic Pseudocyst Drainage
Acronym: ZEUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: M.I.Tech Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Tae Jun Song, MD, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZEUS-PPD-001
Record Dates: First submitted 2025-02-23; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Pseudocyst
Keywords: Pancreatic Pseudocyst; Endosonography; Drainage; Stents
MeSH Terms: conditions — Pancreatic Pseudocyst

STUDY DESIGN:
Intervention Model Description: The design is non-randomized, with no control or comparison group. The study aims to assess both clinical and technical success, as well as device-related safety outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Intervention Group (Experimental): Participants will undergo endoscopic ultrasound-guided drainage of pancreatic pseudocysts using the HANAROSTEN® HOT Plumber™ with Z-EUSIT™.
  Interventions: Device: HANAROSTEN® HOT Plumber™ with Z-EUSIT™

INTERVENTIONS:
Device: HANAROSTEN® HOT Plumber™ with Z-EUSIT™ — An electrocautery-enhanced lumen-apposing metal stent designed for the drainage of pancreatic pseudocysts. The stent is delivered using a system that allows for single-step deployment without the need for guidewire exchanges or tract dilation.

SUMMARY:
The goal of this prospective, single-center observational study is to evaluate the safety and effectiveness of the HANAROSTEN® HOT Plumber™ with Z-EUSIT™ for draining pancreatic pseudocysts.

The main questions the study aims to answer are:

* Does the device reduce the size of pancreatic pseudocysts by at least 50% and improve associated symptoms within 30 to 60 days?
* Can the stent be successfully placed, retained, and removed without complications?

Participants will:

* Undergo endoscopic ultrasound-guided transgastric or transduodenal drainage of pancreatic pseudocysts using the HANAROSTEN® HOT Plumber™ with Z-EUSIT™.
* Be monitored for adverse events such as bleeding, infection, stent migration, or tissue injury.
* Return for follow-up visits within 30 or 60 days for stent removal and evaluation of clinical success.

The study will:

* Enroll 20 adults aged 18 years or older who meet the inclusion criteria.
* Conduct follow-up assessments until one month after stent removal.

DETAILED DESCRIPTION:
Detailed Description

This prospective, single-center observational study aims to evaluate the safety and effectiveness of the HANAROSTEN HOT Plumber with Z-EUSIT for pancreatic pseudocyst drainage. The study will assess clinical success, defined as a reduction of at least 50% in pseudocyst size accompanied by symptom improvement, as well as technical success, device retention, lumen patency, and adverse events. Follow-up will continue until one month after stent removal.

### Study Rationale

* Pancreatic pseudocysts develop due to pancreatic duct obstruction or damage caused by inflammation, resulting in fluid accumulation. Symptoms may include abdominal pain, gastric outlet obstruction, early satiety, and weight loss. Drainage is required when pseudocysts become symptomatic, infected, or increase in size.
* Endoscopic ultrasound-guided transgastric or transduodenal drainage is the standard treatment for accessible pseudocysts. Compared to surgical or percutaneous methods, this approach is less invasive and promotes faster recovery.
* The HANAROSTEN HOT Plumber with Z-EUSIT features an electrocautery-enhanced delivery system, eliminating the need for guidewire exchanges and tract dilation. The stent is made of nitinol wire with silicone coating and anti-migration bi-flanges, designed for easy placement and removal.

Study Design

* Type: Prospective, single-center, observational study
* Device: HANAROSTEN HOT Plumber with Z-EUSIT
* Target Enrollment: 20 adults aged 18 years or older
* Procedure: Endoscopic ultrasound-guided transgastric or transduodenal drainage of pancreatic pseudocysts
* Follow-Up: Until one month after stent removal

Procedure Overview

* Prior to the procedure, cross-sectional imaging (CT or MRI) will determine pseudocyst size and proximity to the gastrointestinal lumen, guiding stent selection.
* Patients will receive prophylactic antibiotics and sedation with midazolam and pethidine according to institutional protocols.
* Under EUS guidance, the pseudocyst will be punctured using the electrocautery-enhanced delivery system. The stent will be deployed to create a connection between the pseudocyst and the gastrointestinal lumen, allowing fluid drainage.
* If direct puncture is not feasible, a 19-gauge needle will be used to access the pseudocyst, followed by guidewire placement and stent deployment.
* Stent removal will occur after pseudocyst resolution, confirmed by follow-up imaging, and will be performed using forceps or a snare.

Follow-Up and Safety Monitoring

* Participants will be monitored for adverse events, including bleeding, infection, perforation, stent migration, tissue injury, and other complications.
* Follow-up visits will occur within 30 or 60 days after the procedure, and one month after stent removal.
* Safety monitoring will include clinical assessments, laboratory tests, and imaging studies as required.

Data Collection and Statistical Analysis

* Data will be summarized using descriptive statistics. Continuous variables will be reported as mean ± standard deviation or median (interquartile range), and categorical variables as frequencies and percentages.
* Technical success rates will be calculated as the percentage of successful stent placements and removals. Clinical success rates will be reported as the percentage of participants with ≥50% pseudocyst size reduction and symptom improvement.
* Adverse events will be classified according to severity and relationship to the device. The incidence of stent migration, retention, and lumen patency will also be reported.
* Missing data will be handled using the last observation carried forward (LOCF) method.

Ethical Considerations

* The study will be conducted in accordance with the Declaration of Helsinki and Good Clinical Practice guidelines.
* All participants will provide written informed consent before enrollment.
* Personal data will be anonymized and securely stored, accessible only to authorized study personnel.

This study aims to provide clinical evidence supporting the safety and effectiveness of the HANAROSTEN HOT Plumber with Z-EUSIT for pancreatic pseudocyst drainage, potentially improving outcomes for patients with this condition.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older
* Diagnosed with pancreatic or peripancreatic pseudocyst or walled-off necrosis (with less than 30% solid components)
* Eligible for endoscopic ultrasound-guided drainage
* Able to provide informed consent and comply with study procedures

Exclusion Criteria:

* Younger than 18 years old
* Pseudocysts with the following characteristics:
* Immature pseudocyst
* Cystic neoplasm
* Pseudoaneurysm
* Multiple pseudocysts requiring drainage
* Uncontrolled coagulation disorders:
* INR > 1.5
* Platelet count < 50,000/mm³
* Other bleeding disorders
* Ineligibility for EUS-guided drainage due to anatomical or technical reasons
* History of anaphylactic reaction to stent materials
* Pregnant or potentially pregnant women
* Current participation in another clinical trial that may affect study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-25 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Success | Within 30 or 60 days after stent placement
  Reduction of pancreatic pseudocyst size by at least 50% with improvement in associated symptoms.

SECONDARY OUTCOMES:
Technical Success - Stent Placement | During procedure
  Successful deployment of the stent at the intended site.
Technical Success - Stent Removal | Within 30 or 60 days after placement
  Successful removal of the stent after pseudocyst resolution, confirmed by endoscopic confirmation of complete stent removal without residual fragments.
Stent Retention | Within 30 or 60 days after placement
  Retention of the stent in the intended location without migration until removal.
Lumen Patency | Within 30 or 60 days after placement
  Maintenance of an open lumen allowing fluid drainage until stent removal.
Procedure Duration | During procedure
  Time from initial needle puncture to full deployment of the stent.
Adverse Events | From procedure day until one month after stent removal
  Incidence of complications such as bleeding, infection, perforation, stent migration, tissue injury, or other adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Dongwook Oh, MD, PhD, Study Director — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional policies and confidentiality regulations.